CLINICAL TRIAL: NCT03899337
Title: A Phase II, Randomised Study of CHOP-R in Combination With Acalabrutinib Compared to CHOP-R in Patients With Newly Diagnosed Richter's Syndrome and a Platform for Initial Investigations Into Activity of Novel Treatments in Relapsed/Refractory and Newly Diagnosed Richter's Syndrome.
Brief Title: A Trial of CHOP-R Therapy, With or Without Acalabrutinib, in Patients With Newly Diagnosed Richter's Syndrome
Acronym: STELLAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Bloodwise (Other); Acerta Pharma, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_17-194
Record Dates: First submitted 2019-03-20; First posted 2019-04-02 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Richter Syndrome
Keywords: Chronic Lymphocytic Leukaemia; Richter's Transformation; Richter's Syndrome; CHOP-R; Acalabrutinib; Diffuse Large B Cell Lymphoma; non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — acalabrutinib; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Standard of Care Arm (CHOP-R) (Active Comparator): Arm in the randomised trial. CHOP-R chemoimmunotherapy will continue for up to 6 cycles (each cycle is 21 days), and will be given according to the following schedule:
  Rituximab, 375 mg/m2, IV infusion, OD, 6 cycles, days of cycle: 1 Cyclophosphamide, 750 mg/m2, IV bolus, OD, 6 cycles, days of cycle: 1 Doxorubicin, 50 mg/m2, IV bolus, OD, 6 cycles, days of cycle: 1 Vincristine, 1.4 mg/m2, IV infusion, OD, 6 cycles, days of cycle: 1 Prednisolone, 40 mg/m2, PO, OD, 6 cycles, days of cycle: 1-5
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: Rituximab
- Experimental Arm (CHOP-R + Acalabrutinib) (Experimental): Arm in the randomised trial. CHOP-R chemoimmunotherapy will continue for up to 6 cycles (each cycle is 21 days), and will be given according to the following schedule:
  Rituximab, 375 mg/m2, IV infusion, OD, 6 cycles, days of cycle: 1 Cyclophosphamide, 750 mg/m2, IV bolus, OD, 6 cycles, days of cycle: 1 Doxorubicin, 50 mg/m2, IV bolus, OD, 6 cycles, days of cycle: 1 Vincristine, 1.4 mg/m2, IV infusion, OD, 6 cycles, days of cycle: 1 Prednisolone, 40 mg/m2, PO, OD, 6 cycles, days of cycle: 1-5
  Acalabrutinib 100 mg, PO, BD will be taken on days 6-21, of each cycle - up to cycle 6. Acalabrutinib treatment will be continuous thereafter until disease progression toxicity, patient choice or death.
  Interventions: Drug: Acalabrutinib; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: Rituximab
- Cohort 1 - Acalabrutinib Monotherapy - Platform Trial (Experimental): Registration arm in platform study. Patients registered to Cohort 1 will receive 100 mg acalabrutinib monotherapy, twice daily, continuously from day 1 until disease progression, toxicity, patient choice or death.
  Interventions: Drug: Acalabrutinib
- Cohort 2 - CHOP-R + Acalabrutinib - Platform Trial (Experimental): Registration arm in platform study. CHOP-R chemoimmunotherapy will continue for up to 6 cycles (each cycle is 21 days), and will be given according to the following schedule:
  Rituximab, 375 mg/m2, IV infusion, OD, 6 cycles, days of cycle: 1 Cyclophosphamide, 750 mg/m2, IV bolus, OD, 6 cycles, days of cycle: 1 Doxorubicin, 50 mg/m2, IV bolus, OD, 6 cycles, days of cycle: 1 Vincristine, 1.4 mg/m2, IV infusion, OD, 6 cycles, days of cycle: 1 Prednisolone, 40 mg/m2, PO, OD, 6 cycles, days of cycle: 1-5
  Acalabrutinib 100 mg, PO, BD will be taken on days 6-21, of each cycle - up to cycle 6. Acalabrutinib treatment will be continuous thereafter until disease progression toxicity, patient choice or death.
  Interventions: Drug: Acalabrutinib; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — 100mg capsule, PO, BD
  Arms: Cohort 1 - Acalabrutinib Monotherapy - Platform Trial; Cohort 2 - CHOP-R + Acalabrutinib - Platform Trial; Experimental Arm (CHOP-R + Acalabrutinib)
Drug: Cyclophosphamide — 750mg/m^2, IV bolus
  Arms: Cohort 2 - CHOP-R + Acalabrutinib - Platform Trial; Experimental Arm (CHOP-R + Acalabrutinib); Standard of Care Arm (CHOP-R)
Drug: Doxorubicin — 50mg/m^2, IV bolus
  Arms: Cohort 2 - CHOP-R + Acalabrutinib - Platform Trial; Experimental Arm (CHOP-R + Acalabrutinib); Standard of Care Arm (CHOP-R)
Drug: Vincristine — 1.4mg/m^2, IV infusion
  Arms: Cohort 2 - CHOP-R + Acalabrutinib - Platform Trial; Experimental Arm (CHOP-R + Acalabrutinib); Standard of Care Arm (CHOP-R)
Drug: Prednisolone — 40mg/m^2, PO, OD
  Other Names: Pevanti
  Arms: Cohort 2 - CHOP-R + Acalabrutinib - Platform Trial; Experimental Arm (CHOP-R + Acalabrutinib); Standard of Care Arm (CHOP-R)
Drug: Rituximab — 375mg/m^2, IV infusion
  Other Names: Mabthera
  Arms: Cohort 2 - CHOP-R + Acalabrutinib - Platform Trial; Experimental Arm (CHOP-R + Acalabrutinib); Standard of Care Arm (CHOP-R)

SUMMARY:
The STELLAR trial will assess the effect of acalabrutinib taken in combination with CHOP-R compared to taking CHOP-R alone in patients with newly diagnosed Richter's Syndrome (RS). It will also be a platform to test other new drugs that show potential for treating RS. Chronic lymphocytic Leukaemia (CLL) is the most common blood cancer in adults, usually in their 70s or older. In a few patients, CLL can transform from a slow-growing cancer into an aggressive lymphoma called Richter's Syndrome. RS is very difficult to treat and patients have a short life-expectancy - usually a few months after diagnosis. Treatment for Richter's Syndrome in the UK is CHOP (four chemotherapy drugs) plus rituximab ('R' - an antibody treatment). The CHOP-R treatment is given as a standard of care for RS but has limited benefit - it is often temporary to extend life. Richter's Syndrome returns in most patients who then die from this disease. The STELLAR trial will investigate if a new drug called acalabrutinib, which is effective used by itself in patients with relapsed CLL and also some with Richter's Syndrome, will improve outcomes for newly diagnosed patients with RS. Acalabrutinib blocks a protein in CLL which can stop the cancer growing.

Participants who have Richter's Syndrome and are suitable for CHOP-R will be recruited by specialised hospitals across the UK. People with another cancer, heart problems, or recent stroke cannot take part. Participants will have a lymph node biopsy, 3-4 bone marrow biopsies, blood samples, and PET-CT and CT scans. CHOP-R is given in a hospital every three weeks up to 6 times. All participants will receive CHOP-R; half will also receive acalabrutinib. When treatment with CHOP-R ends the patients who had acalabrutinib can continue to take it; patients who had CHOP-R alone may have acalabrutinib if their Richter's Syndrome returns after CHOP-R.

DETAILED DESCRIPTION:
Trial Design:

STELLAR is a UK multi-centre trial for patients with newly-diagnosed Richter's Syndrome (RS), which is a rare and highly aggressive transformation of another blood cancer, chronic lymphocytic leukaemia (CLL). It has two parts: a randomised trial (the main component of the trial) which compares the current standard of care with an 'experimental' combination, and a platform for trialing single-arm studies investigating new drugs, or new combinations of drugs, for treating patients with newly-diagnosed Richter's Syndrome. The first novel treatment to be investigated in STELLAR is acalabrutinib which is a 'small molecule' drug that targets and blocks one of the pathways that causes the CLL (and by extension Richter's Syndrome) cancer cells to grow and multiply. Stopping the proliferation of cancer cells is a key aim of cancer treatments. There have been promising studies using acalabrutinib to treat patients with CLL and patients with Richter's Syndrome, but so far these are small and have not compared acalabrutinib, on its own or in a combination, with the current Standard of Care treatment for Richter's Syndrome: CHOP-R chemotherapy (cyclophosphamide, doxorubicin, vincristine, prednisolone and rituximab). In the STELLAR trial we will investigate if adding acalabrutinib to CHOP-R gives a better outcome for patients than CHOP-R alone. The sample sizes described below have been calculated by biostatisticians and are based on the known rates of progression, survival, and response rates for patients with Richter's Syndrome. The sample sizes given below will enable us to answer the research questions with the appropriate number of patients with a strong confidence interval.

In the randomised component of STELLAR, 60 eligible patients will be randomised 1:1 between the current standard of care for Richter's Syndrome (CHOP-R) and the experimental treatment of CHOP-R plus acalabrutinib such that 30 patients are in each of these two sets. The trial is not blinded so participants, clinic staff, and trial staff will know which treatment they receive after the patient has been randomised. Participants will have frequent assessments, which includes assessments after 4 and 6 cycles of treatment to see if the treatment is working, and all patients will be followed up for a minimum of 2 years. The primary aim of the randomised component is to see if adding acalabrutinib to CHOP-R improves the rate of progression free survival (PFS) for RS patients, i.e. if they are in remission from Richter's Syndrome for a longer period of time. It is important that this component is randomised so that the comparison of the two treatments will be fair and unbiased.

In the platform study part of STELLAR, single-arm cohorts (not randomised) will receive treatment which will test the activity of novel combinations or treatment. The platform may be expanded to test other promising treatments if any are identified whilst the randomised trial is open to recruitment. In the first platform study there are two cohorts which will answer two different research questions. The platform arms are not randomised or blinded because they are not comparable; it is rather that they help us to determine whether these treatments may be possible candidates for future therapies.

* Cohort 1 (21-30 participants) will be made up of patients whose Richter's Syndrome has progressed (their disease has got worse) whilst being treated with CHOP-R (or CHOP + another immunotherapy treatment) alone or who have relapsed with Richter's Syndrome after completing treatment with CHOP-R. Entry to this cohort will be prioritised for patients who have taken part in the STELLAR randomised trial, but will be opened up to patients outside STELLAR if fewer than 21 patients from STELLAR take part. In this cohort we will investigate if giving acalabrutinib treatment on its own improves outcomes for patients who have got worse on or relapsed after the current standard of care (CHOP-R).
* Cohort 2 (up to 15 patients) are anthracycline-naïve (they haven't received CHOP-R before) Richter's Syndrome patients, who have been diagnosed whilst being treated with ibrutinib (defined as a diagnosis within 4 weeks of the last dose of ibrutinib). Ibrutinib is the same class of drug as acalabrutinib, though acalabrutinib is a newer drug. Ibrutinib is often used to treat CLL and it is not known if patients who have been treated with ibrutinib will respond to treatment with acalabrutinib if they have Richter's Syndrome. Ibrutinib is becoming a routine treatment for CLL, so it is important to find out if acalabrutinib will help patients who do not respond to ibrutinib. These patients are not included in the randomised trial so that we can determine if acalabrutinib will work in these ibrutinib-treated patients.

Participants:

Participants will be identified at specialist haemato-oncology centres around the UK through multidisciplinary team meetings and consultant referral from other centres. Patients will be approached by their consultant and other, trained, members of the clinic team to introduce and discuss the trial. Patients will receive a patient information sheet and will be given at least 24 hours to review the information and ask any additional questions they may have.

Patients who have enrolled on STELLAR who are offered entry into Cohort 1 because their disease has worsened when treated with CHOP-R alone, will already be familiar with the trial processes and systems. They will need to know all of the new information about acalabrutinib (the treatment for Cohort 1) and will be provided with a separate patient information sheet, clinicians will aim to give patients at least 24 hours to review the information. Because these patients are already familiar with the trial and will need urgent treatment they may be permitted to consent on the same day that they have received the patient information sheet if they have all their questions answered and are happy to proceed.

Treatment:

Participants randomised to the standard of care arm will receive up to 6 cycles of CHOP-R where each cycle is 21 days. Participants will be treated in a hospital day unit on day 1 of each cycle and will have tablets to take at home on days 2 to 5. All participants will be formally assessed after 4 and 6 cycles of treatment. Participants who have achieved a response may continue on to a stem cell transplant if they are suitable. Participants who do not achieve a response will be offered entry in to the platform Cohort 1 to receive acalabrutinib monotherapy if they are eligible. Entry into Cohort 1 is not mandatory; the participant's doctor will discuss all possible treatment options with them.

Participants who consent and are registered to Cohort 1 will take 100 mg twice-daily of acalabrutinib at home as oral tablets. Treatment is continuous until disease progression, unacceptable toxicity or patient choice. Participants will be formally assessed at weeks 12 and 24 to determine if they are responding to treatment.

Participants randomised to the experimental arm of STELLAR and registered to Cohort 2 will receive up to 6 cycles of CHOP-R where each cycle is 21 days. Participants will be treated in a hospital day unit on day 1 of each cycle and will have tablets to take at home on days 2 to 5. Patients will then take 100 mg twice daily of acalabrutinib oral tablets at home on days 6-21. All participants will be formally assessed after 4 and 6 cycles of treatment. Participants who have achieved a response will continue to take acalabrutinib at home at 100 mg twice daily, continuously until disease progression, unacceptable toxicity or patient choice. These participants may continue on to a stem cell transplant if they are suitable. If these patients do not achieve a response, they will discontinue trial treatment.

In all cases, if patients do not respond to treatment or wish to withdraw from the trial they will be counselled by their medical team on the options available to them.

Assessments and visits:

Participants in the STELLAR trial will have frequent assessments in the first 4 to 6 months of the study so that they are monitored for toxicity and response to treatment. Most of the assessments for participants receiving CHOP-R (with or without acalabrutinib) would be done as part of their standard of care. Before entering the study each potential participant will undergo screening assessments in the 4 weeks before trial entry (date of randomisation or registration).

Screening assessments:

A physical and medical assessment by their doctor to record their: age, medical history, blood pressure, pulse, weight, any symptoms of their Richter's Syndrome, ECG (heart trace), and any other relevant information. Women who are could become pregnant have to have a pregnancy test. Blood samples are taken for local assessments (blood count and other haematology tests, biochemistry, virology, immunology) and also for research (these are 'extra' samples that are not standard of care). Patients will also have a bone marrow assessment, a PET-CT scan, and a lymph node biopsy; these assessments would be done as part of the patients' standard of care.

Assessments during the trial:

All patients will have local assessments carried out whilst they receive CHOP-R, most of these assessments are standard of care. Patients will have extra assessments that will help us to answer the exploratory questions posed in the trial. Most of these extra assessments will be done at the same time as local assessments so that patients don't have lots of extra visits to the hospital. Patients in all cohorts will have: a physical assessment by their doctor to record their blood pressure, pulse, weight, and any symptoms or side effects they may have; blood samples are taken for local assessments, patients receiving acalabrutinib will have more blood samples taken for research at the same time as the local ones.

All patients will have a lymph node biopsy, bone marrow biopsy and PET-CT scan as part of their screening assessments. Some patients may have a bone marrow biopsy at the end of cycle 6 (or week 24 for Cohort 1) which would be part of their standard of care. All patients will have a CT scan at the end of cycle 4 (week 12 for Cohort 1) and a PET-CT at the end of cycle 6 (week 24 for Cohort 1). If a patient has disease progression they will have another PET-CT scan and lymph node biopsy, and some patients will have a bone marrow biopsy. All of these scans and biopsies would be part of the patient's standard of care.

As well as medical assessments, patients will complete validated Quality of Life questionnaires at trials visits. There are three multi item scales on fatigue, treatment side effects and disease symptoms, infection and social activities and future health worries. These questionnaires will be completed at clinic visits.

Follow Up:

All STELLAR patients will be followed-up for disease status and survival for at least 2 years from trial entry to determine the long-term effectiveness of the therapy.

ELIGIBILITY:
Entry criteria for randomised trial component (standard of care and experimental arms):

Inclusion criteria for the randomised trial component:

* Suitable for anthracycline-containing chemo-immunotherapy.
* Patients with CLL and newly diagnosed biopsy proven DLBCL-type RS.
* ECOG performance status of 0, 1, 2 or 3.
* Age 16 years and over.
* Signed written informed consent prior to performing any study-specific procedures.

Exclusion criteria for the randomised trial component:

* Prior therapy with CHOP or any anthracycline containing treatment at any time prior to randomisation. (Please note that pre-treatment with prednisolone up to 2mg/kg is allowed for up to 14 days prior to the start of treatment).
* Ibrutinib-exposed CLL patients who have been newly diagnosed with RS within four weeks of their last dose of ibrutinib. (Ibrutinib-exposed CLL patients who discontinue ibrutinib due to toxicity or progressive CLL and later (more than four weeks) develop RS are not excluded from the randomised trial component).
* Previous acalabrutinib exposure. (Prior exposure to other Bruton tyrosine kinase (BTK), phosphoinositide-3-kinase (PI3K), or BCL-2 inhibitors is permitted, with the exception of patients who have progressed on ibrutinib - see exclusion criterion above).
* Known central nervous system (CNS) involvement of CLL or DLBCL.
* Any other active malignancy that requires active treatment, with the exception of basal cell carcinoma, in-situ cervical cancer, and non-invasive squamous cell carcinoma of the skin.
* Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, and active hepatitis
* Positive serology for Hepatitis B (HB) defined as a positive test for HB surface antigen (HBsAg). In addition, if negative for HBsAg but HB core antibody (HBcAb) positive (regardless of HBsAb status), a HBV deoxyribonucleic acid (DNA) test will be performed and if positive the patient will be excluded.
* Known human immunodeficiency virus (HIV) positive.
* Patients with active bleeding or history of bleeding diathesis (e.g. haemophilia, von Willebrand disease).
* Patients receiving therapeutic anticoagulation with warfarin or equivalent (e.g. phenprocoumon).
* Uncorrected prolonged prothrombin time (PT) or an activated partial thromboplastin time (APTT) > 2 x the upper limit of normal (ULN).
* Major surgery within 30 days prior to randomisation and/or inadequate recovery (at Investigators discretion) from any prior major surgery, toxicity or complications.
* Patients with malabsorption syndrome or medical conditions significantly affecting gastrointestinal function.
* Clinically significant cardiac disease including unstable angina, uncontrolled congestive heart failure, and unstable arrhythmias requiring therapy, with the exception of extra systoles or minor conduction abnormalities. Stable and controlled atrial fibrillation is not an exclusion.
* Significant concurrent, uncontrolled severe medical condition including, but not limited to, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease.
* History of significant cerebrovascular disease in the 6 months prior to randomisation, including intracranial haemorrhage.
* Known or suspected hypersensitivity to components of the investigational products
* Patients who have received treatment with any non-marketed drug substance or experimental therapy within 4 weeks prior to proposed start of treatment unless discussed and approved by the Chief Investigator or Clinical Coordinator via the Trials Office.
* Current participation in any other interventional clinical study.
* Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder).
* Breast feeding women or women with a positive pregnancy test at screening.
* Women of childbearing potential and men not willing to use highly effective contraception during study and for 12 months after last dose of study therapy. Highly effective contraception is defined as abstinence, hormonal birth control, intrauterine devices, vasectomy/surgical sterilisation.

Entry criteria for single-arm relapsed Cohort 1:

Inclusion criteria for Cohort 1 (progressive RS following chemo-immunotherapy):

* Patients with relapsed/refractory RS who received anthracycline based chemotherapy with anti-CD20 monoclonal antibody If fewer than the expected number of patients from the randomised component enter into Cohort 1, patients from outside STELLAR with relapsed/refractory RS following chemo-immunotherapy (anthracycline based chemotherapy with anti-CD20 monoclonal antibody) will be able to join this cohort if they meet the eligibility criteria. The Trials Office will alert sites by email if any slots are released for patients outside of STELLAR, these must be booked with the Trials Office prior to registration.
* ECOG performance status of 0, 1, 2 or 3.
* Age 16 years and over.
* Signed written informed consent prior to performing any study-specific procedures.

Exclusion criteria for Cohort 1 (progressive RS following chemo-immunotherapy):

* Previous acalabrutinib exposure. (Prior exposure to other Bruton tyrosine kinase (BTK), phosphoinositide-3-kinase (PI3K), or BCL-2 inhibitors is permitted).
* Known central nervous system (CNS) involvement of CLL or DLBCL.
* Any other active malignancy that requires active treatment, with the exception of basal cell carcinoma, in-situ cervical cancer, and non-invasive squamous cell carcinoma of the skin.
* Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, and active hepatitis
* Positive serology for Hepatitis B (HB) defined as a positive test for HB surface antigen (HBsAg). In addition, if negative for HBsAg but HB core antibody (HBcAb) positive (regardless of HBsAb status), a HBV deoxyribonucleic acid (DNA) test will be performed and if positive the patient will be excluded.
* Known human immunodeficiency virus (HIV) positive.
* Patients with active bleeding or history of bleeding diathesis (e.g. haemophilia, von Willebrand disease).
* Patients receiving therapeutic anticoagulation with warfarin or equivalent (e.g. phenprocoumon).
* Uncorrected prolonged prothrombin time (PT) or an activated partial thromboplastin time (APTT) > 2 x the upper limit of normal (ULN).
* Major surgery within 30 days prior to registration and/or inadequate recovery (at Investigators discretion) from any prior major surgery, toxicity or complications.
* Patients with malabsorption syndrome or medical conditions significantly affecting gastrointestinal function.
* Clinically significant cardiac disease including unstable angina, uncontrolled congestive heart failure, and unstable arrhythmias requiring therapy, with the exception of extra systoles or minor conduction abnormalities. Stable and controlled atrial fibrillation is not an exclusion.
* Significant concurrent, uncontrolled severe medical condition including, but not limited to, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease.
* History of significant cerebrovascular disease in the 6 months prior to registration, including intracranial haemorrhage.
* Known or suspected hypersensitivity to components of the investigational products
* Patients who have received treatment with any non-marketed drug substance or experimental therapy within 4 weeks prior to proposed start of treatment unless discussed and approved by the Chief Investigator or Clinical Coordinator via the Trials Office.
* Current participation in any other interventional clinical study.
* Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder).
* Breast feeding women or women with a positive pregnancy test at screening.
* Women of childbearing potential and men not willing to use highly effective contraception during study and for 12 months after last dose of study therapy. Highly effective contraception is defined as abstinence, hormonal birth control, intrauterine devices, vasectomy/surgical sterilisation.

Entry criteria for single arm Cohort 2

Inclusion criteria for Cohort 2 (anthracycline-naïve RS patients, diagnosed while on ibrutinib):

* Ibrutinib-exposed CLL patients who have developed biopsy-proven DLBCL-type RS within four weeks of last dose of ibrutinib.
* No previous anthracycline treatment and suitable for anthracycline-containing chemo-immunotherapy.
* Patients with CLL and newly diagnosed biopsy proven DLBCL-type RS.
* ECOG performance status of 0, 1, 2 or 3.
* Age 16 years and over.
* Signed written informed consent prior to performing any study-specific procedures.

Exclusion criteria for Cohort 2 (anthracycline-naïve RS patients, diagnosed while on ibrutinib):

* Prior therapy with CHOP or any anthracycline containing treatment at any time prior to registration. (Please note that pre-treatment with prednisolone up to 2mg/kg is allowed for up to 14 days prior to the start of treatment).
* Previous acalabrutinib exposure. (Prior exposure to other Bruton tyrosine kinase (BTK), phosphoinositide-3-kinase (PI3K), or BCL-2 inhibitors is permitted)
* Known central nervous system (CNS) involvement of CLL or DLBCL.
* Any other active malignancy that requires active treatment, with the exception of basal cell carcinoma, in-situ cervical cancer, and non-invasive squamous cell carcinoma of the skin.
* Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, and active hepatitis
* Positive serology for Hepatitis B (HB) defined as a positive test for HB surface antigen (HBsAg). In addition, if negative for HBsAg but HB core antibody (HBcAb) positive (regardless of HBsAb status), a HBV deoxyribonucleic acid (DNA) test will be performed and if positive the patient will be excluded.
* Known human immunodeficiency virus (HIV) positive.
* Patients with active bleeding or history of bleeding diathesis (e.g. haemophilia, von Willebrand disease).
* Patients receiving therapeutic anticoagulation with warfarin or equivalent (e.g. phenprocoumon).
* Uncorrected prolonged prothrombin time (PT) or an activated partial thromboplastin time (APTT) > 2 x the upper limit of normal (ULN).
* Major surgery within 30 days prior to registration and/or inadequate recovery (at Investigators discretion) from any prior major surgery, toxicity or complications.
* Patients with malabsorption syndrome or medical conditions significantly affecting gastrointestinal function.
* Clinically significant cardiac disease including unstable angina, uncontrolled congestive heart failure, and unstable arrhythmias requiring therapy, with the exception of extra systoles or minor conduction abnormalities. Stable and controlled atrial fibrillation is not an exclusion.
* Significant concurrent, uncontrolled severe medical condition including, but not limited to, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease.
* History of significant cerebrovascular disease in the 6 months prior to registration, including intracranial haemorrhage.
* Known or suspected hypersensitivity to components of the investigational products
* Patients who have received treatment with any non-marketed drug substance or experimental therapy within 4 weeks prior to proposed start of treatment unless discussed and approved by the Chief Investigator or Clinical Coordinator via the Trials Office.
* Current participation in any other interventional clinical study.
* Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder).
* Breast feeding women or women with a positive pregnancy test at screening.
* Women of childbearing potential and men not willing to use highly effective contraception during study and for 12 months after last dose of study therapy. Highly effective contraception is defined as abstinence, hormonal birth control, intrauterine devices, vasectomy/surgical sterilisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Randomised Component - Progression free survival (PFS) | Time from randomisation to the date of progression or death from any cause, whichever came first, assessed up to 24 months..
  Progression free survival (PFS) defined as the time from randomisation to the date of progression or death from any cause. Progression will be defined by the modified Cheson criteria (Appendix 1). Patients who are alive and progression free at the time of analysis will be censored at date last seen. Any participants who withdraw or are lost to follow-up will also be censored at date last seen.
Registration Arm - Cohort 1 - Overall Response | Response assessed at 24 weeks of treatment
  Overall response after 24 weeks of treatment based on the modified Cheson criteria (Appendix 1). Complete response (CR) and partial response (PR) are considered to be positive responses for assessment of this outcome. Participants who withdraw prior to the 6 month assessment or do not have the 6 month assessment will be considered non responders.
Registration Arm - Cohort 2 - Overall Response | Response assessed after 6 cycles of treatment. Each cycle is 21 days.
  Overall response after 6 cycles of treatment, defined by the modified Cheson criteria (Appendix 1). CR and PR are considered to be positive responses for assessment of this outcome. Participants who withdraw prior to the post-cycle-6 assessment or do not have the post-cycle-6 assessment will be considered non-responders.

SECONDARY OUTCOMES:
Overall Survival | Time from trial entry to the date of death from any cause, whichever came first, assessed up to 24 months.
  Defined as time from date of randomisation (for randomised trial) or registration (to the relevant cohort for single-arm cohorts) to date of death from any cause.
  Participants who are alive at the time of analysis will be censored at date last seen.
Overall Response after 6 cycles | Response assessed after 6 cycles of treatment. Each cycle is 21 days.
  Overall response (randomised component only) after cycle 6, defined by the modified Cheson criteria (Appendix 1). CR and PR are considered to be positive responses for assessment of this outcome. Participants who withdraw prior to the post-cycle-6 assessment or do not have the post-cycle-6 assessment will be considered non-responders.
Overall Response after 12 weeks | Response assessed after 12 weeks of treatment
  Overall response (cohorts 1 only) after 12 weeks, defined by the modified Cheson criteria (Appendix 1). CR and PR are considered to be positive responses for assessment of this outcome. Participants who withdraw prior to the 12-week assessment or do not have the 12- week assessment will be considered non-responders.
Progression Free Survival | Time from date of registration to date of progression or death from any cause, whichever came first, assessed up to 24 months.
  PFS (single-arm cohorts only) defined as the time from date of registration to date of progression or death from any cause. Progression will be defined by the modified Cheson criteria (Appendix 1). Participants who are alive and progression free at the time of analysis will be censored at date last seen. Any patients who withdraw or are lost to follow-up will also be censored at date last seen.
Quality of Life Questionnaire Outcomes | Analysed at the end of cycles 4 (week 12) and 6 (week 24)
  QoL, (assessed using ECOG performance status [Appendix 7]), and the CLL17 and NHLHG29 questionnaires (Appendix 2)) at the end of cycles 4 and 6 for participants receiving CHOP-R as part of their treatment (randomised cohorts and Cohort 2), and at 12 and 24 weeks for participants receiving acalabrutinib monotherapy (Cohort 1).
Exhibited Toxicity | Measured from start of treatment until 28 days after last dose
  Toxicity defined as the number of participants who experience one or more adverse event grade 3 or higher or serious adverse event of any grade.
Proportion of patients proceeding to allogeneic or autologous stem cell transplantation | Confirmation of partial or complete remission, assessed at the following time points: Randomised Trial/ Platform Study - Cohort 2: Post Cycle 4, Post Cycle 6 (where each cycle is 21 days); Platform Study - Cohort 1: Week 12, Week 24.
  Measured as proportion of patients proceeding to transplant on each treatment arm, at confirmation of partial or complete remission

CONTACTS AND LOCATIONS:
Overall Officials: Anna Schuh, PhD, Principal Investigator — University of Oxford
Locations (16):
- United Kingdom (16):
  - Belfast City Hospital, Belfast
  - Royal Bournemouth Hospital, Bournemouth
  - University Hospital of Wales, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - King's College Hospital, London
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Christie Hospital, Manchester
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klintman J, Appleby N, Stamatopoulos B, Ridout K, Eyre TA, Robbe P, Pascua LL, Knight SJL, Dreau H, Cabes M, Popitsch N, Ehinger M, Martin-Subero JI, Campo E, Mansson R, Rossi D, Taylor JC, Vavoulis DV, Schuh A. Genomic and transcriptomic correlates of Richter transformation in chronic lymphocytic leukemia. Blood. 2021 May 20;137(20):2800-2816. doi: 10.1182/blood.2020005650. PMID 33206936
- [Derived] Appleby N, Eyre TA, Cabes M, Jackson A, Boucher R, Yates F, Fox S, Rawstron A, Hillmen P, Schuh A. The STELLAR trial protocol: a prospective multicentre trial for Richter's syndrome consisting of a randomised trial investigation CHOP-R with or without acalabrutinib for newly diagnosed RS and a single-arm platform study for evaluation of novel agents in relapsed disease. BMC Cancer. 2019 May 20;19(1):471. doi: 10.1186/s12885-019-5717-y. PMID 31109313